CLINICAL TRIAL: NCT03470051
Title: A Prospective Multi-center Case Collection Study of Breast Imaging Examinations From Women With Non-suspicious Breast Masses to Correlate the Calculated Mass Doubling Time Using Quantitative Transmission Ultrasound (QT Ultrasound) With Mass Histology.
Brief Title: Case Collection Study in the Evaluation of Doubling Time Rates in Non-Suspicious Breast Masses Using QT Ultrasound Technology
Acronym: EVALUATE
Status: Completed | Type: Observational
Sponsor: QT Ultrasound LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BR007
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- (2) QT Ultrasound scans prior to breast biopsy: Subjects will undergo a baseline QT scan, and a follow-up QT scan performed between 90 days and 180 days from their baseline QT Scan accompanied by a HHUS and ultrasound-guided breast biopsy following the first follow-up QT scan. BI-RADS will be confirmed by the radiologist at the time of the first HHUS. Subjects will receive a telephone follow-up contact approximately 2-3 business days after their ultrasound-guided breast biopsy to assess if any adverse events have occurred. Subjects will be asked to come back for an additional follow-up QT Scan 12 months from the time of their baseline QT Scan.
  Interventions: Diagnostic Test: QT Ultrasound
- (0-1) QT Ultrasound scans prior to breast biopsy: Subjects that have not had (2) two QT Scans before their breast biopsy and who haven't yet had a breast biopsy will undergo an optional baseline QT scan accompanied by a HHUS and ultrasound-guided breast biopsy. BI-RADS will be confirmed by the radiologist. Subjects will receive a telephone follow-up contact approximately 2-3 business days after their ultrasound-guided breast biopsy to assess if any adverse events have occurred. Subjects will be asked to come back for a follow-up QT Scan between 90 and 180 days from the time of their study biopsy.
  Subjects that have had a breast biopsy on their identified breast mass(es) prior to study enrollment and have not already had two (2) QT Scans will undergo an optional baseline QT scan if between 0 and 30 days from their breast biopsy.
  Subjects will be asked to come back for a follow-up QT Scan 12 months from the time of their study biopsy.
  Interventions: Diagnostic Test: QT Ultrasound

INTERVENTIONS:
Diagnostic Test: QT Ultrasound — All subjects will be asked to agree to an ultrasound-guided breast needle biopsy by a qualified radiologist experienced in this procedure if not already completed prior to study entry.

SUMMARY:
This is a prospective case collection study to collect cases for subsequent statistical studies and future reader studies.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18 or older
3. Willing to receive QT Ultrasound Breast Scans
4. Willing to undergo an ultrasound-guided needle breast biopsy if performed after enrollment in the study
5. Willing and able to provide Informed Consent prior to any research-related procedure(s)
6. Have an identified solid non-suspicious breast mass

Exclusion Criteria:

1. Pregnancy
2. Currently breastfeeding
3. Magnetic material in the chest which in the judgement of the Principal Investigator would interfere or be impacted by the magnets utilized with the study device.
4. Not willing to provide information for primary care physician
5. History of breast cancer
6. History of treated or untreated cancer of a non-breast origin which in the judgment of the Principal Investigator would be a concern for metastatic disease to the breast
7. Physical inability to tolerate the QT scan, i.e. inability to lie prone and still for up to 30 minutes at a time
8. Open wounds, sores or skin rash present on the breast(s) or nipple discharge from the scanned breast(s)
9. Breasts too large for scanner, i.e. bra size larger than DDD or inability to successfully "fit" breast after the subject is placed on scanner
10. Body weight greater than 400 lbs. (180 kg)
11. Concurrent disease or condition which in the judgment of the Principal Investigator disqualifies the subject from participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects must be female
Study Population: Subjects with a non-suspicious breast mass will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Breast mass doubling time change | 90 days
  The change in calculated mass doubling time using Quantitative Transmission Ultrasound (QT Ultrasound) from a minimum of two study timepoints will be measured and compared to mass histology.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Memorial Care Long Beach, Long Beach, California
  - Marin Breast Health Trial Center, Novato, California

IPD SHARING:
Plan to Share IPD: No